CLINICAL TRIAL: NCT06480604
Title: A Pilot Clinical Trial Assessing the Effect of a Multi-strain Probiotic on the Risk of Recurrence and Severity of Symptoms in Females With Recurrent Vulvovaginal Candidiasis
Brief Title: Effect of a Multi-strain Probiotic on Recurrent Vulvovaginal Candidiasis
Acronym: PROVELIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CTB2022TN202
Record Dates: First submitted 2024-06-25; First posted 2024-06-28 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Microbiome; Probiotic; Recurrent; Vulvovaginal; Candidiasis; RVVC; Vaginal; Chronic; Infection
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Recurrence; Candidiasis; Bronchiolitis Obliterans Syndrome; Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants in this arm will receive a daily dose of 2x10^9 Colony Forming Units (CFU) of a multi strain probiotic (live bacterium), corresponding to 2 capsules once daily, for 6 months.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants in this arm will receive an equivalent placebo for the duration of the study (6 months).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants in this arm will receive a daily dose of 2x10^9 Colony Forming Units (CFU) of a multi strain probiotic (live bacterium), corresponding to 2 capsules once daily, for 6 months.
  Arms: Probiotic
Dietary Supplement: Placebo — Participants in this arm will receive an equivalent placebo for the duration of the study (6 months).
  Arms: Placebo

SUMMARY:
This study evaluates the effect of a multi-strain probiotic on the risk of recurrence and severity of symptoms in females with recurrent vulvovaginal candidiasis (R-VVC).

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of live bacteria on the incidence and severity of symptoms of vulvovaginal candidiasis (VVC) recurrence. The trial will be run in India and recruit women with recurrent vulvovaginal candidiasis (R-VVC).

ELIGIBILITY:
Inclusion Criteria:

Individuals meeting ALL of the following criteria will be enrolled for the study:

1. Premenopausal women aged 18-50 years.
2. Women with a culture-confirmed active episode caused by Candida spp. (albicans or non-albicans) reported within 24-48 hours of evidence of clinical symptoms. (No medications should have been initiated before the sample for culture is collected).
3. Documented history of recurrence of at least 3 VVC episodes in the last 12 months confirmed by vaginal culture /clinical diagnosis.
4. Culture growth of Candida spp. causing VVC.
5. Random Capillary Blood Glucose of < 110mg/dl.
6. Willingness to consume the study products for the entire study duration.
7. Willing to complete all study procedures and comply with study requirements.
8. Willing to abstain from other supplements or medication.
9. Ready to give voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

Individuals meeting ANY of the following criteria will be excluded from the study:

1. Post-menopausal and peri-menopausal women.
2. Pregnant/breast-feeding women.
3. Use of oral or vaginal anti-fungal medication in the last 14 days.
4. Vaginal culture suggestive of bacterial vaginosis (Nugent's score of 7-10), trichomonas vaginalis or Gardnerella vaginalis.
5. Participants found positive for Clotrimazole resistance, by vaginal culture & sensitivity at screening.
6. Known allergy to Clotrimazole.
7. Women not willing to use any form of vaginal medication during the study.
8. Use of vaginal douching.
9. Unwillingness to use an appropriate method of contraception.
10. Diagnosed with compromised immune system, type I and/or type II diabetes mellitus, or malignancies.
11. Use of corticosteroids therapy in the last 30 days.
12. Use of oral/systemic antimicrobial therapy in the last 30 days.
13. Known allergy to the study products or azoles.
14. Individuals with a history of frequent infections requiring antibiotic treatments.
15. Participation in another clinical study(ies) in the last 3 months.
16. Women who, in the opinion of the Investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the study.
17. Women with uncontrolled hypertension with systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg.
18. Heavy alcohol drinkers defined as follows: For men, consuming more than 4 drinks on any day or more than 14 drinks/week. For women, consuming more than 3 drinks on any day or more than 7 drinks/week.
19. Smokers.
20. History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders that, in the judgment of the Investigator, would interfere with the participant's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the individual at undue risk.
21. Presence of unstable, acutely symptomatic, or life-limiting illness.
22. Use of any supplements (includes probiotics, post-biotics, herbal supplements, synbiotics, enzyme supplements, vitamins with probiotics) in the last 30 days.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal women aged 18-50 years, with a culture-confirmed active VVC episode caused by Candida spp. (albicans or non-albicans) and reported within 24-48 hours of evidence of clinical symptoms.
Enrollment: 126 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of culture-confirmed VVC recurrence between baseline and day 180 as compared to placebo. | Day 0, Day 180
  Efficacy of a multi-strain probiotic on incidence of culture-confirmed VVC recurrence as compared to placebo, where VVC recurrence is defined as a fungal culture positive vaginal swab with at least 2 moderate VVC related symptoms or at least 1 severe VVC related symptom and with VVC free period prior to this incident of at least 7 days.

SECONDARY OUTCOMES:
Occurrence of culture-confirmed VVC recurrence between baseline and day 90 as compared to placebo. | Day 0, Day 90
  Efficacy of a multi-strain probiotic on incidence of culture-confirmed VVC recurrence as compared to placebo, where VVC recurrence is defined as a fungal culture positive vaginal swab with at least 2 moderate VVC related symptoms or at least 1 severe VVC related symptom and with VVC free period prior to this incident of at least 7 days.
Time to first recurrence of VVC episode from baseline between probiotic and placebo groups. | Day 0 to first VVC recurrence
  Time to first recurrence of VVC episode from baseline between probiotic and placebo groups, where VVC recurrence is defined as a fungal culture positive vaginal swab with at least 2 moderate VVC related symptoms or at least 1 severe VVC related symptom and with VVC free period prior to this incident of at least 7 days.
Change in the number of days with VVC episode between probiotic and placebo groups. | Duration (days) of VVC episodes, Day 0-180.
  Efficacy of a multi-strain probiotic on the number of days with VVC episode as compared to placebo group, where VVC episode is defined as a fungal culture positive vaginal swab with at least 2 moderate VVC related symptoms or at least 1 severe VVC related symptom and with VVC free period prior to this incident of at least 7 days.
Change in severity of VVC episodes between probiotic and placebo groups. | During VVC episodes
  Efficacy of a multi-strain probiotic on the severity of VVC episodes as assessed by symptoms (itching/soreness, edema, dysuria, vaginal discharge, dyspareunia, erythema, fissures/excoriations) severity on a 4-point Likert Scale as compared to baseline and placebo.
  The number of days of an episode will be captured using the e-dairy. First day of the episode will be considered as the day when the participant experiences onset of at least 2 moderate symptoms or at least one severe symptom on the 4-point Likert scale. The last day of the episode will be considered when there is no presence of VVC related clinical signs and symptoms and thus the composite score on the Likert scale is 0.
Proportion of Candida albicans positive VVC episodes vs other pathogens between probiotic and placebo groups. | During VVC episodes
  Efficacy of a multi-strain probiotic on proportion of Candida albicans positive VVC episodes vs other pathogens.
Number of administrations of vaginal pessaries during acute VVC episodes as compared to baseline and placebo. | During VVC episodes
  Number of vaginal pessaries applied during acute VVC episodes as compared to baseline and placebo. A Clotrimazole 100 mg pessary to be applied once daily at bedtime till no symptoms persist.
Changes in vaginal health as assessed by vaginal pH and compared to baseline and placebo. | Day 0, Day 90, Day 180
  Changes in vaginal health as assessed by vaginal pH, compared to baseline and placebo, using pH strips.
Changes in vaginal microbiology as assessed by vaginal Candida albicans culture and compared to baseline and placebo. | During episodes
  Changes in vaginal microbiology as assessed by vaginal Candida albicans culture and compared to baseline and placebo.
Quality of life as assessed using SF-36 and compared to baseline and placebo. | Day 0, Day 90, Day 180
  Changes in quality of life as assessed using SF-36 and compared to baseline and placebo.
  Total and individual scoring of the 8 sections of the SF-36 questionnaire will be used to infer the improvement in quality of life improve. A high score defines a more favorable health state (maximum score 100).

OTHER OUTCOMES:
Influence of multi-strain probiotic on vaginal microbiome as compared to baseline and placebo. | Day 0, Day 90, Day 180
  Effects of a multi-strain probiotic in vaginal microbiome as assessed by shotgun analysis and compared to baseline and placebo.

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - Anand Multispeciality Hospital, Vadodara, Gujarat
  - Life Care Hospital, Nashik, Maharashtra
  - AMF's Moraya Multispeciality Hospital, Pune, Maharashtra
  - ENT & Vertigo Clinic, Pune, Maharashtra
  - Vivaan Hospital, Sopāra, Maharashtra
  - Matritva Women's Hospital, Vasai, Maharashtra

IPD SHARING:
Plan to Share IPD: No